CLINICAL TRIAL: NCT00420615
Title: An Open Label Phase I Study to Evaluate the Effects of Patupilone on the Pharmacokinetics of Midazolam and Omeprazole in Patients With Advanced Malignancies
Brief Title: Evaluate the Effects of Patupilone on the Pharmacokinetics of Midazolam and Omeprazole in Patients With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CEPO906A2123
Record Dates: First submitted 2007-01-10; First posted 2007-01-11 (Estimated); Last update posted 2020-12-08 (Actual); Status verified 2012-04

CONDITIONS: Solid Tumors
Keywords: Cancer; EPO906; Patupilone
MeSH Terms: conditions — Neoplasms | interventions — epothilone B; Omeprazole

ARMS (2):
- Patupilone and Omeprazole (Experimental): patupiloe + omeprazole
  Interventions: Drug: Patupilone and Omeprazole
- patupilone + midalzolam (Experimental): patupilone + midalzolam
  Interventions: Drug: Patupilone + Midalzolam

INTERVENTIONS:
Drug: Patupilone and Omeprazole
  Arms: Patupilone and Omeprazole
Drug: Patupilone + Midalzolam
  Arms: patupilone + midalzolam

SUMMARY:
The purpose of this study is to evaluate the potential inhibitory effects of patupilone on metabolism using midazolam and omeprazole as the respective probe drugs.

ELIGIBILITY:
Inclusion criteria:

* Male or female patients 18 years or older
* Histologically documented advanced solid tumor, who have failed standard systemic therapy, or for whom standard systemic therapy does not exist
* Life expectancy of 3 months or more
* Patients with adequate hematologic parameters

Exclusion criteria:

* Hypersensitivity to midazolam or omeprazole or related compounds
* Female patients who are pregnant or breast-feeding.
* Patients with a severe and/or uncontrolled medical disease
* Patients with a known diagnosis of human immunodeficiency virus (HIV) infection
* Patients having received an investigational agent within 30 days prior to study entry

Other protocol defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2006-12; Primary Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the effects of patupilone on the pharmacokinetics of midazolam in patients with advanced malignancies. | Day 1 (0.5h, 1h, 1.5h, 3h, 4h, 6h, 8h, 12h, 24h, 36h, 48h), Day 29 (0.5h, 1h, 1.5h, 3h, 4h, 6h, 8h, 12h, 24h, 36h, 48h)
To evaluate the effects of patupilone on the pharmacokinetics of omeprazole in patients with advanced malignancies | Day 1 (0.33h (20m), 0.67h (40m), 1h, 1.5h, 2h, 2.5h, 3h, 4h, 6h, 8h, 10h, 12h)

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of Patupilone when administered concomitantly with midazolam in patients with advanced malignancies. | at each visit (week 1, week 2, week 5, and end of study)
To evaluate the safety and tolerability of Patupilone when administered concomitantly with omeprazole in patients with advanced malignancies. | at each visit (week 1, week 2, week 5, and end of study)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmeceuticals
Locations (1):
- The University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: Results can be found for CEPO906A2123 on the Novartis Clinical Trials Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=6803